CLINICAL TRIAL: NCT04115176
Title: Smoking Effects on GCF GCF IL-17A AND IL-17 Levels and Oxidative Status of Patients Receiving Periodontal Treatment
Brief Title: GCF IL-17 Levels and Oxidative Status of Smoking and Non-smoking Individuals With Periodontitis
Acronym: GCF
Status: Completed | Type: Observational
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, muge lutfioglu, Associate Professor, Ondokuz Mayıs University
Other Study IDs: PYO.DIS.1901.17.002
Record Dates: First submitted 2019-10-02; First posted 2019-10-03 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Chronic Periodontitis; Smoking, Cigarette
Keywords: chronic periodontitis; smoking,; periodontal treatment,; IL-17,; oxidative stress
MeSH Terms: conditions — Chronic Periodontitis; Cigarette Smoking; Smoking

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- smokers + periodontitis: Individuals clinically diagnosed with chronic periodontitis that smoke recruited for this group.
- nonsmoker + periodontitis: Individuals clinically diagnosed with chronic periodontitis that don't smoke recruited for this group.

SUMMARY:
This study was performed to evaluate the effects of both periodontal treatment and smoking on the gingival crevicular fluid(GCF) levels of interleukin (IL)-17A, IL-17E, Total oxidative stress(TOS) and total antioxidant capasity(TAOC) in smoking and non-smoking patients with severe chronic periodontitis.

Systemically healthy 15 smoker,15 non-smoker with chronic periodontitis were attended for the study. Periodontal status were determined by recording periodontal clinical measurements. GCF samples were collected at the baseline, at the end of initial periodontal treatment and 4 weeks after periodontal flap surgery. The data were tested statistically by the Student t and paired sample t tests.

ELIGIBILITY:
Inclusion Criteria:

* individuals aged ˃35 years and having ≥16 teeth diagnosed as chronic periodontitis
* not received any periodontal therapy within the previous 6 months;
* not received antibiotic/anti-inflammatory drug treatment within the previous 6 months.

Exclusion Criteria:

* receiving medical treatment for cancer, rheumatoid arthritis, diabetes mellitus, cardiovascular disease, or any other systemic disease;
* being pregnant or being in the period of menopause or lactation;
* receiving any drug therapy that might affect the clinical characteristics of periodontitis;
* usage of systemic antimicrobials during the 6 weeks prior to data collection

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with chronic periodontitis (with an age range of 35 to 60 years) seeking dental treatment at the Periodontology Clinic, School of Dentistry, Ondokuz Mayis University, were included in the present study.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2019-07-10 (Actual); Study Completion 2019-07-10 (Actual)

PRIMARY OUTCOMES:
GCF IL-17A VOLUME | GCF sampling was performed prior to periodontal treatment , 4 weeks after completion of initial periodontal treatment, and 4 weeks after periodontal flap surgery .
  IL-17A is a cytokine present in gingival crevicular fluid. Its volume calculated as microliter and changes due to inflammation caused by periodontal disease.
GCF IL-17E VOLUME | GCF sampling was performed prior to periodontal treatment , 4 weeks after completion of initial periodontal treatment, and 4 weeks after periodontal flap surgery .
  IL-17E is a cytokine present in gingival crevicular fluid. Its volume calculated as microliter and changes due to inflammation caused by periodontal disease.
GCF TOTAL OXIDATIVE STRESS (TOS) LEVEL | GCF sampling was performed prior to periodontal treatment , 4 weeks after completion of initial periodontal treatment, and 4 weeks after periodontal flap surgery .
  TOS is the measurement of oxidative stress amount and given as mmol/L unit. Its amount changes due to inflammation caused by periodontal disease.
GCF TOTAL ANTIOXIDANT CAPASITY (TAOC) | GCF sampling was performed prior to periodontal treatment , 4 weeks after completion of initial periodontal treatment, and 4 weeks after periodontal flap surgery .
  TAOC is the antioxidant amount measured and given as μmol H2O2 Eq/L unit. Its amount changes due to inflammation caused by periodontal disease.

CONTACTS AND LOCATIONS:
Overall Officials: MÜGE LÜTFİOĞLU, Principal Investigator — assoc. prof.
Locations (1):
- Müge Lütfioğlu, Samsun, Atakum, Turkey (Türkiye)